CLINICAL TRIAL: NCT07403760
Title: Wellbeing and Survival Improvement With Event Reduction by Ablation for Atrial Fibrillation in the Very Elderly (WISER-AF)
Brief Title: Wellbeing and Survival Improvement With Event Reduction by Ablation for Atrial Fibrillation in the Very Elderly
Acronym: WISER-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS202607
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: catheter ablation; very elderly; quality of life
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter Ablation Group (Experimental)
  Interventions: Procedure: Catheter Ablation
- Sham Control Group (Sham Comparator)
  Interventions: Procedure: Sham Control

INTERVENTIONS:
Procedure: Catheter Ablation — Patients undergo PVI (for paroxysmal AF) or PVI +linear ablation+EI-VOM(for persistent AF) using pulsed field ablation catheters. All patients will wear eye masks and headphones with music during the procedure.
  Arms: Catheter Ablation Group
Procedure: Sham Control — Patients undergo femoral vein puncture and catheter placement. Phrenic nerve stimulation is performed to mimic procedural sensations. No ablation energy is delivered. All patients will wear eye masks and headphones with music during the procedure. Patients remain in the lab for at least 80 minutes.
  Arms: Sham Control Group

SUMMARY:
The WISER-AF trial is a multicenter, double-blind, sham-controlled, randomized controlled trial. It aims to evaluate the efficacy and safety of catheter ablation compared to a sham procedure in improving the quality of life (SF-36 score) in very elderly patients (aged ≥80 years) with symptomatic atrial fibrillation over a 6-month follow-up period.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) prevalence increases with age, posing significant challenges in the very elderly (≥80 years). While catheter ablation is an established treatment for general AF patients, its efficacy in improving quality of life (QoL) in the very elderly remains underrepresented in previous trials. The WISER-AF trial is designed to fill this evidence gap. The study will enroll 182 symptomatic AF patients aged ≥80 years in China. Patients will be randomized 1:1 to undergo either pulsed field ablation (PFA) or a sham procedure. To ensure blinding, all patients will wear eye masks and headphones during the procedure. The sham group will receive phrenic nerve stimulation to mimic the sensation of ablation without delivering therapeutic energy. The primary endpoint is the change in the SF-36 total score from baseline to 6 months. Secondary endpoints include changes in AFEQT score, Clinical Frailty Scale (CFS), LVEF, NT-proBNP, 6-minute walk distance, and cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 80 years.
2. Documented paroxysmal or persistent atrial fibrillation by ECG or Holter within 6 months prior to enrollment.
3. Symptomatic AF (including palpitations, chest tightness, fatigue, dizziness, blackouts, dyspnea).
4. Voluntary participation and signed informed consent.

Exclusion Criteria:

1. NYHA Class IV heart failure.
2. Acute myocardial infarction, cardiac surgery, or PCI within the past 1 year.
3. Long-standing persistent AF (duration > 1 year).
4. Left atrial anteroposterior diameter > 6 cm.
5. History of prior AF ablation.
6. AF secondary to reversible causes (e.g., post-surgery, infection, hyperthyroidism).
7. Severe mitral stenosis.
8. Moderate to severe hepatic failure (Child-Pugh B-C).
9. Renal failure stage 4-5 (eGFR <30 ml/min/1.73m2) or continuous dialysis.
10. Inability to cooperate due to dementia or severe mental disorder.
11. Presence of left atrial thrombus.
12. Prior Left Atrial Appendage Occlusion (LAAO).
13. Contraindication to anticoagulation.
14. Life expectancy < 1 year.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in SF-36 Total Score | Baseline, 6 months
  Difference in the change of the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) total score from baseline to 6 months between the two groups.

SECONDARY OUTCOMES:
Change in AFEQT Score | Baseline, 6 months
  Change in Atrial Fibrillation Effect on Quality-of-Life (AFEQT) score
Change in Clinical Frailty Scale (CFS) Score | Baseline, 6 months
  Change in frailty status assessed by CFS
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline, 6 months
Change in NT-proBNP level | Baseline, 6 months
Change in 6-Minute Walk Distance (6MWT) | Baseline, 6 months
Freedom from Atrial Arrhythmias | 6 months
  Absence of atrial fibrillation, atrial flutter, or atrial tachycardia recorded by ECG, Holter, or patch monitor after a 30-day blanking period.
Incidence of Composite Cardiovascular Outcome | 6 months
  Composite of all-cause death, stroke or systemic embolism, myocardial infarction, major bleeding, and heart failure hospitalization/emergency visits.
Healthcare Resource Utilization | 6 months
  Number of emergency room visits and unplanned hospitalizations
Serious Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Prof., Principal Investigator — Beijing Anzhen Hospital; Ning Zhou, Prof., Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China, Beijing, China

IPD SHARING:
Plan to Share IPD: No